CLINICAL TRIAL: NCT02979132
Title: Evaluation of the Validity of a Novel Isotope Dilution Method to Assess the Iron Status and Its Changes in Swiss Women
Brief Title: Iron Long-Term Labelling Study Switzerland
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prof. Michael B. Zimmermann (Other)
Responsible Party: Sponsor-Investigator, Prof. Michael B. Zimmermann, Professor, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Fe_LTL_Swi
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Iron Absorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Iron Supplementation (Active Comparator): Eisensulfat LOMAPHARM 50 mg administration for 90 days
  Interventions: Drug: Eisensulfat LOMAPHARM 50 mg
- Intravenous Iron Supplementation (Active Comparator): Single-dose Ferinject(R) administration
  Interventions: Drug: Ferinject(R)
- Food Fortification with Iron (Active Comparator): Consumption of iron-fortified biscuits (15 mg Fe in form of FeSO4) for 90 d
  Interventions: Dietary Supplement: iron fortified biscuits

INTERVENTIONS:
Drug: Eisensulfat LOMAPHARM 50 mg — oral intake of an 'Eisensulfat LOMAPHARM 50 mg' tablet every morning for 90 days
  Other Names: Eisentabletten
  Arms: Oral Iron Supplementation
Drug: Ferinject(R) — Single-dose Ferinject(R) administration
  Other Names: Iron Infusion
  Arms: Intravenous Iron Supplementation
Dietary Supplement: iron fortified biscuits — consumption of an iron-fortfied biscuit every morning for 90 days
  Other Names: HUG-Biskuits
  Arms: Food Fortification with Iron

SUMMARY:
Conventional indirect indicators of iron status, using serum and red blood cell biomarkers, are confounded by inflammation from common infections and are therefore of limited use in populations carrying a high burden of infection and inflammation, as for example women of reproductive age in malaria endemic areas in developing countries. Even without the confounding effect of inflammation, current markers of iron status are insensitive to small changes in dietary iron and do not allow to establish associations between dietary, lifestyle and genetic factors and iron balance. With a new method based on the dilution of a previously administered and equilibrated stable isotope signal, an accurate measurement of long-term oral iron balance and absorption is possible, allowing the estimation of iron requirements and potentially providing fundamental guidance for supplementation and fortification programs in both healthy and chronically inflamed/infected patients. In the current study the novel methodology will be validated in generally healthy subjects with low iron status. The technique will be used to assess dietary and lifestyle determinants of iron status and to compare the effect on iron balance and iron status of three distinct, commonly used iron interventions: food fortification with iron; oral iron supplementation, and intravenous iron infusion.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in a former absorption study in our lab,
* Signed written informed consent to participate in the new study,
* Serum ferritin < 25 µg/L

Exclusion Criteria:

* Anaemia (Hb < 117 g/L),
* Any metabolic, gastrointestinal, kidney or chronic disease such as diabetes, renal failure, hepatic dysfunction, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement),
* Allergic or similar reactions against iron supplements,
* Known fructose intolerance, glucose-galactose malabsorption or saccharase-isomaltase deficiency,
* Known hypersensitivity to ponceau R4 and ponceau R4 aluminium salt (E124)
* Continuous/long-term use of medication during the whole study (except for contraceptives),
* Regular consumption of mineral and vitamin supplements within 2 weeks prior to 1st supplement administration (more than 3 consecutive days or more than 5 times within 14 days),
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 6 months,
* pregnancy or breast feeding,
* Intention to become pregnant during the course of the study,
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Enrollment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
iron isotope composition in blood | 9 months
  tracer to tracee rate in venous blood samples at different time points

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Laboratory, ETH Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Speich C, Mitchikpe CES, Cercamondi CI, Zeder C, Brittenham GM, Moretti D, Zimmermann MB. Direct assessment of body iron balance in women with and without iron supplementation using a long-term isotope dilution method in Benin and Switzerland. Am J Clin Nutr. 2021 Jun 1;113(6):1657-1669. doi: 10.1093/ajcn/nqaa433. PMID 33693464